CLINICAL TRIAL: NCT04308928
Title: Evaluation of New Biomarker-based Approaches for Improving the Diagnosis of Childhood Tuberculous Meningitis
Acronym: TBMBIOMARKER
Status: Completed | Type: Observational
Sponsor: University of Stellenbosch (Other)
Collaborators: European and Developing Countries Clinical Trials Partnership (EDCTP) (Other Government); Medical Research Council, South Africa (Other)
Responsible Party: Principal Investigator, Novel Njweipi Chegou, Principal Investigator, University of Stellenbosch
Other Study IDs: UStellenboschTBM
Record Dates: First submitted 2020-03-11; First posted 2020-03-16 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Tuberculous Meningitis
Keywords: Tuberculosis; meningitis; childhood tuberculous meningitis
MeSH Terms: conditions — Tuberculosis, Meningeal; Tuberculosis; Meningitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Cerebrospinal fluid, serum, urine
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Children with suspected meningitis: Patients must have a clinical diagnosis of meningitis including one or more of the following symptoms: headache, irritability, vomiting, fever and neck stiffness (Table 1). The diagnosis of probable or possible TBM is based on 1) clinical findings 2) CSF results 3) neuroimaging findings 4) evidence for TB outside the central nervous system and 5) additional laboratory criteria. A scoring system then determines whether a patient falls in the probable or possible TBM category. Points are allocated for a positive finding in each of the categories, with a maximum score for each category. A total score of at least 10 is compatible with probable TBM, while a total score of at least 6 equates with a possible TBM diagnosis.
- Children with definite tuberculous meningitis: Definite TBM requires demonstration of acid- fast bacilli in the CSF, Mycobacterium tuberculosis culture from CSF, a positive nucleic acid amplification test (PCR) of CSF or histopathological evidence of Mycobacterium tuberculosis from a central nervous system site.

SUMMARY:
The rapid diagnosis of tuberculosis (TB) in children remains a serious challenge owing to limitations in the existing diagnostic tests. TB meningitis (TBM), an extrapulmonary form of TB, is the most severe manifestation of paediatric TB. TBM results in high morbidity and mortality in children, despite the availability of chemotherapy, mainly due to diagnostic delay. Most tests required for proper TBM diagnosis including analysis of cerebrospinal fluid (CSF) and brain imaging are not available in resource-limited settings e.g., in most of Africa including South Africa. New tests for TBM are urgently needed. The main goal of this proposal is to develop a point-of-care (POC) diagnostic test for TBM, based on CSF and bloodbiomarkers.

Aim 1: Evaluate the diagnostic potentials of 51 host inflammatory biomarkers that the investigators recently identified in CSF and blood samples from children with suspected meningitis in a repository of 100 stored CSF and serum samples using a multiplex platform. After statistical analysis including multi-marker modelling by linear discriminant analysis, random forest, and other modelling techniques, the investigators will select the best combination of up to four biomarkers for incorporation into the prototype diagnostic test (Aim 2).

Aim 2: Incorporate the best performing CSF and serum biomarkers into a novel, patented biosensor-based POC diagnostic test. The investigators will develop a multi-biomarker prototype test for detecting up to 4 biomarkers in serum or CSF.

Aim 3: Evaluate the newly developed POC test on 300 children prospectively. This will be done at the Tygerberg Academic Hospital. The diagnostic yield of the POC test will be compared to the routine diagnostic tests.

DETAILED DESCRIPTION:
Introduction:

te ongoing research, early and cost-effective diagnostic tools for TBM are lacking. The detection of Mycobacterium tuberculosis (Mtb) in cerebrospinal fluid (CSF) is the gold standard for diagnosing TBM. Unfortunately the sensitivity of both smear microscopy and culture for TBM is low. Depending on the reference standard employed, the sensitivity of the GeneXpert test (Cepheid Inc, USA) for TBM is approximately 50-60%, and improved to 72% when centrifuged CSF was used in one study. In a more recently published study conducted on HIV positive adults, however, the GeneXpert performed with a sensitivity of 43% or 45%, compared to 43% or 45% for culture and 70% or 95% for the GeneXpert Ultra, depending on which of the two reference standards were used. Despite the relatively high roll-out of the GeneXpert test across South Africa, the test is currently mostly offered at centralised laboratories. The availability of the test in other African countries is limited. The diagnosis of TB relies on the poorly sensitive symptom screening and smear microscopy, especially at rural health centres. Mtb culture facilities are often only available at referral level laboratories and results might take up to 42 days. The need for multiple health care visits leads to loss of follow-up and delayed diagnosis, fuelling the spread of TB and advanced lung damage. In the case of TBM in particular, proper diagnosis is only made upon admission in a tertiary level referral center. In routine clinical practice, diagnosis is mostly based on a combination of clinical findings, multiple laboratory tests on the CSF, imaging findings and the exclusion of common differential diagnoses. Most of these techniques are unavailable in many high-burden, but resource-constrained settings in most of sub-Saharan Africa. Children seen at primary and secondary healthcare facilities often have multiple missed opportunities, up to six visits, before eventual diagnosis of TBM is made in a relatively well-resourced setting in South Africa. Findings from the CSF can be highly variable. Recently, international experts have proposed new uniform case definitions that should be employed in future research to replace the many different definitions in the literature. New tests are therefore urgently needed for the diagnosis of TBM.

The investigators investigated the potential of host markers detected in CSF samples from children suspected of having TBM as diagnostic candidates for TBM . The investigators evaluated the levels of the host biomarkers present in a standard BioPlex 27plex multiplex cytokine kit (Bio Rad Laboratories) and other protein biomarkers in CSF and serum samples. An unsupervised hierarchical clustering and principal component analysis, using the Glucore Omics explorer, revealed significant clustering of patients with TBM by the biomarkers detected in the CSF. A 3-marker host protein biosignature comprising vascular endothelial growth factor (VEGF), interleukin (IL)-13 and the antibacterial peptide cathelicidin, LL-37, showed potential as a diagnostic biosignature for TBM (international patent application: PCT/IB2015/052751), diagnosing TBM with an area under the receiver operator characteristics curve (AUC) of 0.91, with sensitivity of 52%, but with good specificity of 95%. Since the publication of this biosignature, the investigators have evaluated the diagnostic potential of >70 host biomarkers in serum and plasma samples from adults suspected of having active pulmonary TB in 5 different African countries (South Africa, Namibia, Malawi, Uganda and Ethiopia) in an EDCTP-funded trial (AE-TBC). The investigators identified, patented (PCT/IB2015/051435 and PCT/IB2017/052142), and published 6- and 7-marker protein biosignatures with strong diagnostic potential for TB.

In a more recent study (South African Provisional Patent application; Manyelo et al 2019), the investigators hypothesized that at least some of the host biomarkers comprising our adult protein biosignatures may be useful for TBM diagnostics. Funded by the South African Technology Innovation Agency (PI: Chegou), the investigators prospectively enrolled a new cohort of children suspected of having TBM at the Tygerberg Academic Hospital, Western Cape, and determined the concentrations of 66 host biomarkers, in CSF samples from these children. The investigators also included the 3 biomarkers that comprised our previous CSF biosignature for TBM (VEGF, IL-13 and cathelicidin LL-37) for validation purposes in this new study; a total of 69 host protein biomarkers.

With the exception of VEGF (AUC of 0.81), the accuracy of the individual markers in the previous 3-marker signature was poor (AUCs of 0.58 and 0.55, respectively, for IL-13 and LL-37) but when used in combination the discrimination between TBM and no-TBM by the 3-marker model was confirmed [AUC of 0.67 (95% CI: 0.52-0.83); sensitivity of 75% and specificity of 65%]. Forty-seven of the additional markers showed significant differences between the TBM and no TBM groups (Mann Whitney U test), with 28 showing strong diagnostic potential, even as individual markers (AUC ≥ 0.80). These markers include interferon (IFN)-γ, CCL18(MIP-4), CXCL9, CCL1, CCL5(RANTES), IL-6, tumour necrosis factor (TNF)-α, myeloperoxidase (MPO), matrix metalloproteinase 9 (MMP), MMP-8, complement C2 (CC2), IL-10, total plasminogen activator inhibitor 1 (PAI-1), CXCL8, IL-1β, alpha-2-antitrypsin(A1AT), CXCL10, granulocyte colony stimulating factor (G-CSF), CC4, CC4b, granulocyte-macrophage colony stimulating factor (GM-CSF), platelet-derived growth factor (PDGF)-AB/BB, apolipoprotein A1 (apoA1), mannose-binding lectin (MBL), ferritin, CC5a, serum amyloid P (SAP), and CC5.

Combinations of these biomarkers were investigated and using Linear Discriminant Analysis (LDA) models. A 4-marker CSF biosignature comprising soluble intracellular adhesion molecule (sICAM)-1, MPO, CXCL8 and IFN-γ diagnosed TBM with an AUC of 0.97 (95% CI: 0.92-1.00), with a sensitivity of 87% (20/23) and specificity of 95.8% (23/24). After leave-one-out cross validation, there was no change in the sensitivity and specificity of the 4-marker biosignature. Further optimization of the 4-marker biosignature by the selection of better cut-off values resulted in a sensitivity and specificity of 96% and 96%, respectively.

As VEGF performed well in single-marker analyses (19), the investigators evaluated the potential accuracy of other biosignatures that included VEGF. A 3-marker model comprising VEGF, IFN-γ and MPO discriminated with high accuracy between the children with and without TBM. In leave-one-out cross validation and optimizations of best cut-off values, the sensitivity and specificity of the 3-marker VEGF-based signature were 92% and 100%, respectively.

All 69 host markers investigated in CSF samples were also investigated on serum samples using the Luminex multiplex platform. The median serum levels of 17 analytes [sVCAM1, CCL2, IL-4, TNF-α, CCL4, adipsin, SAP, CC5, CFH, G-CSF, IL-10, Apo-CIII, IL-17A, PAI-1(total), PDGF AB/BB, MBL and NCAM1] were significantly different (p<0.05; Mann Whitney U test) between children with and without TBM. When the diagnostic potential of individual serum biomarkers was assessed by ROC curve analysis, 13 of the markers had promising AUC ≥ 0.70. LDA demonstrated that optimal diagnosis of TBM was achieved using 3 markers. The most accurate 3-marker serum biosignature for the diagnosis of TBM [adipsin (complement factor D), Ab42 and IL-10] diagnosed TBM with an AUC of 0.84 (95% CI: 0.73-0.96), a sensitivity of 82.6% (19/23) and specificity of 75% (18/24). In leave-one-out cross validation, the sensitivity remained 82.6% (19/23) with the specificity decreasing to 70.3% (17/24). Further optimisation of the biosignature by selection of better cut-off values resulted in an improved sensitivity and specificity of 83% and 83%, respectively.

OVERALL OBJECTIVE The main objective is to validate previously identified host serum and CSF biomarkers and to develop a biosensor-based POC test for the diagnosis of TBM, based on these biomarkers.

The investigators propose to identify a panel of correlated biomarkers that showed potential in previous studies. This will be done to identify biomarkers which can be substituted with each other as the transition from a laboratory-based technological platform such as Luminex to a POC test using a biosensor-based technology is likely to be faced by the loss of some of the markers due to technical reasons or due to unavailability of some of the markers due to antibody ownership or cost issues. Highly correla-ted markers can then substitute such markers. The investigators will test which set of biomarkers works best in the POC diagnostic test platform. Finally, the investigators will evaluate the prototype test prospectively in a new cohort of 300 study participants with suspected TBM as described below.

The prototype test will be based on the best biosignature of CSF or serum biomarkers, depending on which performs best. However, developing the test based on serum biomarkers may be advantageous as CSF samples are difficult to collect. Furthermore, a test based on serum biomarkers may be easily converted to a fingerprick based test, which will be much easier to implement in resource-constrained settings. The investigators are currently evaluating a fingerprick screening test for adult TB based on host biomarkers discovered and validated in serum samples as part of an EDCTP2-funded consortium (www.screen-tb.eu).

ELIGIBILITY:
Inclusion Criteria:

* Children between the ages of 3 months and 13 years with suspected meningitis, and who require CSF examination for routine diagnostic purposes at Tygerberg Children's Hospital.
* Written informed consent will be obtained from parents for inclusion of children 3 months to 7 years old in the study.
* If possible, assent will be obtained in those children older than 7 years who have a normal level of consciousness, i.e. a Glasgow Coma Score (GCS) of 15/15.

Exclusion Criteria:

* Children 13 years and older will be excluded from the study.
* Failure to obtain written consent will also exclude children from the study.

Ages: 3 Months to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: The study will be conducted at Tygerberg Children's Hospital, Parow Valley, Cape Town. The hospital is the tertiary academic hospital of the Faculty of Medicine and Health Sciences, University of Stellenbosch. Children with tuberculous meningitis are referred from primary care day hospitals, district and secondary level hospitals from our drainage area. Children with suspected TBM are referred to our institution to establish the diagnosis of TBM and to treat the complications associated with advanced disease (stage 2 and 3 TBM, e.g. hydrocephalus). Research samples collected for the purposes of the current study shall be processed at the Stellenbosch University Immunology Research Group (SUN-IRG) laboratory, Department of Biomedical Sciences, Faculty of Medicine and Health Sciences.
Sampling Method: Non-Probability Sample
Enrollment: 332 (Actual)
Dates: Start 2020-04-01 (Actual); Primary Completion 2024-10-31 (Actual); Study Completion 2025-07-31 (Actual)

PRIMARY OUTCOMES:
Identify CSF or blood-based biosignatures for the diagnosis of TBM in children | 2019-2021
  We have identified a total of 51 inflammatory biomarkers in CSF and/or serum samples in children with suspected TBM. 47 of these host markers (including 10 of the 14 that showed potential in serum either as individual markers or as part of 3-marker signatures) were detected in CSF samples, with only four of these proteins (CCL2, IL-4, adipsin and Ab42) showing potential only in serum samples. Using a repository of 100 CSF and serum samples, currently available in our biobank, from children with suspected TBM, n=50 with TBM, we will look for correlated markers that can be substituted to identify the best performing biomarker set for the POC device (Aim 2).
Develop a prototype POC diagnostic test platform based on the biosignatures. | 2020-2022
  The validated, best performing CSF and serum biomarkers (sub aims 1a and b) will be incorporated into our POC diagnostic platform, at the Engineering Faculty, SU. The first prototype of the biosensor-based assay was shown to quantify antibodies in bodily fluids in the range of 50 ng/ml - 1 µg/ml (22). We will develop a multibiomarker prototype test for 4 biomarkers in CSF or serum. The prototype multi-biomarker test will undergo prospective evaluation in the field (Aim 3), in years 4 and 5. Assay development will be led by Distinguished Professor Willem Perold, a co-investigator on the project, who will be the lead supervisor of one MSc.Engineering student, with Dr. Chegou as co-supervisor.
Evaluate the newly developed test in a new patient cohort. | 2023-2024
  We will evaluate the newly developed test prospectively in a new cohort of children with suspected TBM.
  Clinical study design Recruitment of study participants will follow a longitudinal cohort design. Children suspected of having meningitis will be recruited and assessed for TBM at Tygerberg Academic Hospital, a tertiary level referral hospital and a teaching hospital for SU. It is the second-largest hospital in South Africa. These children will later be classified as having "definite", "probable", "possible" and "no TBM" based on international, standardized criteria (26).

CONTACTS AND LOCATIONS:
Overall Officials: Novel Chegou, Prof, Principal Investigator — University of Stellenbosch
Locations (1):
- Stellenbosch University Immunology Research Group, Cape Town, Western Cape, South Africa

IPD SHARING:
Plan to Share IPD: No
Participant information will be secured using unique participant ID's (PIDs). Participants are minors, and thus published data will use de-identified participant results.

REFERENCES:
- [Result] Kim D, Perold WJ, Chegou NN. Development of a Biosensor for the Early Detection of Tuberculous Meningitis in Infants. Engineering Proceedings. 2025; 109(1):12. https://doi.org/10.3390/engproc2025109012
- [Result] Manyelo CM, Solomons RS, Snyders CI, Kidd M, Kooblal Y, Leukes VN, Claassen C, Roos K, Stanley K, Walzl G, Chegou NN; TBMBIOMARKERS study group. Validation of host cerebrospinal fluid protein biomarkers for early diagnosis of tuberculous meningitis in children: a replication and new biosignature discovery study. Biomarkers. 2022 Sep;27(6):549-561. doi: 10.1080/1354750X.2022.2071991. Epub 2022 May 12. PMID 35506251
- See also: This website provides information about the study, results and also lists publications from the project. — https://www.su.ac.za/en/faculties/medicine/departments/biomedical-sciences/immunology/edctp-funded-studies

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-04-21): https://cdn.clinicaltrials.gov/large-docs/28/NCT04308928/Prot_SAP_000.pdf